CLINICAL TRIAL: NCT03290508
Title: Long-Term Prospective Registry to Evaluate Treatment Decisions and Clinical Outcomes in Patients With Favorable Intermediate-Risk Localized Prostate Cancer Following Cell Cycle Progression (CCP) Testing (Prolaris® Test)
Brief Title: Long-term Study to Evaluate and Clinical Outcomes in Patients With Favorable Intermediate Risk Localized Prostate Cancer
Status: Terminated | Type: Observational
Why Stopped: There is sufficient follow-up data to meet the endpoints of the study.
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: URO-008
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: Prolaris; Prostate Cancer; Cell Cycle Progression Test
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples With DNA — Formalin-fixed paraffin-embedded (FFPE) tissue from blocks or slides of prostatic adenocarcinoma biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prolaris Testing: Recently diagnosed treatment-naïve patients with early stage localized prostate cancer who undergo Prolaris testing
  Interventions: Diagnostic Test: Prolaris Testing
- No Prolaris Testing: Patients with newly diagnosed favorable intermediate-risk localized prostate cancer who DO NOT undergo Prolaris testing

INTERVENTIONS:
Diagnostic Test: Prolaris Testing — Recently diagnosed treatment-naïve patients with early stage localized prostate cancer who undergo Prolaris testing
  Other Names: RNA expression signature of cell cycle progression genes
  Groups: Prolaris Testing

SUMMARY:
This is a long-term prospective registry study to determine whether Prolaris testing in patients with favorable intermediate risk prostate cancer influences physician management decisions toward conservative treatment in patients with Prolaris low-risk scores without negatively impacting patient oncologic outcomes, thereby sparing low-risk patients from unnecessary treatments and associated side-effects.

DETAILED DESCRIPTION:
This is a long-term prospective registry to evaluate the impact of Prolaris testing on therapeutic decisions in patients with newly diagnosed favorable intermediate-risk localized prostate cancer and to summarize clinical oncologic outcomes. The design of the study is non-interventional, and therefore the protocol will not require a specific treatment plan for study participants. However, in the absence of a universally accepted timeframe for repeat biopsies within existing active surveillance recommendations, study sites will be encouraged to monitor patients for disease progression as per the standard of care (e.g., current National Comprehensive Cancer Network [NCCN] guidelines) with the expectation of a repeat biopsy within 18 months of the initial biopsy.

Patients who undergo Prolaris testing will be included in the registry as well as patients who do not undergo Prolaris testing. Data collection for the first primary objective extends over a 3-year period. During this time, data is collected on the treatment initiated, any follow-up prostate biopsy performed in patients initially treated with active surveillance, definitive treatments performed (with pathology data if surgical therapy is performed), and the reasons definitive treatment was pursued, as well as data related to disease progression such as biochemical recurrence, development of prostate cancer metastases, or disease specific death.

Data collection for the second primary objective extends out to 8 years. During this time data is collected on any follow-up prostate biopsy in patients still treated with active surveillance, definitive treatments performed (with pathology data if surgical therapy is performed), and the reasons definitive treatment was pursued, as well as data related to disease progression such as biochemical recurrence, development of prostate cancer metastases, or disease specific death.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone CCP testing and patients who have not undergone CCP testing will be considered for enrollment in the study.

  1. Willing to provide written informed consent.
  2. Males ≥65 years old.
  3. Newly diagnosed (≤6 months), treatment-naïve patient with histologically proven localized adenocarcinoma of prostate whose initial treatment has not been decided.
  4. Candidate for and considering AS and yet would be eligible for definitive therapy.
  5. Favorable intermediate-risk disease, defined by the NCCN as follows:

     * predominant Gleason grade 3; AND
     * percentage of positive cores <50%; AND
     * no more than 1 of the following NCCN intermediate-risk factors:

       * Gleason grade 7
       * T2b-T2c
       * PSA 10-20 ng/mL
  6. Estimated life expectancy ≥10 years.
  7. Can be monitored for disease progression according to standard of care (e.g., current NCCN guidelines).

Exclusion Criteria:

* 1. Clinical evidence of metastasis or lymph node involvement.
* 2. Received pelvic radiation prior to biopsy.
* 3. Received androgen deprivation therapy (ADT) prior to biopsy; however, 5 alpha-reductase inhibitors (5-ARIs) are permitted.
* 4. Participation in interventional clinical trials.
* 5. Patient is considering watchful waiting.
* 6. Has a known history of hypogonadism.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Newly diagnosed (≤ 6 months), treatment-naïve patients with favorable intermediate-risk localized prostate cancer whose initial treatment has not been decided and who are being seen at Medicare Certification and Training Registry (CTR) practices in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Low Prolaris Score, on Active Surveillance | 3 years
  Proportion of patients with low Prolaris scores who are initially treated with active surveillance
Low Prolaris Score, Definitive Treatment Following Active Surveillance | 3 years
  Proportion of patients with low Prolaris scores and initially treated with active surveillance who proceed to definitive treatment at 3 year follow-up
Low Prolaris Score, Disease Progression Following Delayed Definitive Treatment | 8 years
  Proportion of patients with low Prolaris scores and initially treated with active surveillance and later proceed to definitive treatment who develop disease progression at 5 years subsequent to the start of definitive treatment.

SECONDARY OUTCOMES:
Low Prolaris Score, Time to Definitive Treatment following Active Surveillance | 8 years
  Time to definitive treatment in patients with low Prolaris scores who are initially treated with active surveillance.
No Prolaris Score, on Active Surveillance | 3 years
  Proportion of patients without Prolaris testing who are initially treated with active surveillance.
No Prolaris Score, Definitive Treatment Following Active Surveillance | 3 years
  Proportion of patients without Prolaris testing initially treated with active surveillance who proceed to definitive treatment at 3 year follow-up.
No Prolaris Score, Time to Definitive Treatment Following Active Surveillance | 8 years
  Time to definitive treatment in patients without Prolaris testing who are initially treated with Active Surveillance.
No Prolaris Score, Disease Progression Following Delayed Definitive Treatment | 8 years
  Proportion of patients without Prolaris testing and initially treated with active surveillance who proceed with definitive treatment that develop disease progression at 5 years subsequent to the start of definitive treatment.

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Urology Centers of Alabama, Homewood, Alabama
  - East Valley Urology Center, Mesa, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Arkansas Urology, Little Rock, Arkansas
  - Pacific Urology, Concord, California
  - VA Long Beach Healthcare, Long Beach, California
  - UCI Medical Center, Orange, California
  - Ssg Md Apc, San Jose, California
  - Advanced Urology Institute, Daytona Beach, Florida
  - Urology Group of Florida, Delray Beach, Florida
  - Pinellas Urology, St. Petersburg, Florida
  - 21st Century Oncology, Sunrise, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - North Idaho Urology, Coeur d'Alene, Idaho
  - URO Partners, Westchester, Illinois
  - Wichita Urology, Wichita, Kansas
  - Regional Urology, Shreveport, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Department of Urologic Oncology, Ann Arbor, Michigan
  - Comprehensive Urology, Royal Oak, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - UroLogic, Tupelo, Mississippi
  - Premier Urology Group, LLC, Cranford, New Jersey
  - Premier Urology, Cranford, New Jersey
  - Urologic Research and Consulting LLC, Englewood, New Jersey
  - Stony Brook University, Stony Brook, New York
  - A.M.P. Radiation Oncology, Syracuse, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Carolina Urology Partners, West Columbia, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Rio Grande Urology, El Paso, Texas
  - Seattle Urology Research Center, Burien, Washington

IPD SHARING:
Plan to Share IPD: Yes
Results of Prolaris testing to be shared with patient and patient's provider. Individual participant data will be shared with investigators. Aggregate clinical date will be presented in manuscript form.
Time Frame: Within 1 year of last study out.